CLINICAL TRIAL: NCT04181112
Title: Fecal Microbiota Transplantation (FMT) for Intestinal Decolonization of Multidrug-resistant Opportunistic Pathogens
Brief Title: Fecal Transplant for MDRO Decolonization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Amee Manges, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-00782 FMT.MDRO.RCT.1
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Multi-antibiotic Resistance
Keywords: Fecal Microbiota Transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fecal microbiota transplantation (Experimental)
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)
- Fecal microbiota transplantation with antibiotic pre-treatment (Experimental)
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)
- No intervention follow-up (No Intervention)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — FMT using retention enema
  Arms: Fecal microbiota transplantation; Fecal microbiota transplantation with antibiotic pre-treatment

SUMMARY:
This is a trial designed to determine whether fecal microbiota transplantation (FMT) can eliminate highly drug-resistant bacteria from the intestinal tract of renal transplant patients. The primary goal of this study is to test whether oral gut decontamination followed by FMT using enema delivery will result in decolonization of the intestinal tract of renal transplant patients shortly after solid organ transplantation, thereby preventing difficult to treat post-transplant infections.

DETAILED DESCRIPTION:
Contact the study principal investigator for the study protocol.

ELIGIBILITY:
Renal transplant patient inclusion criteria:

* 18 years or older
* Able to provide informed consent
* Positive for one of the target MDRO by rectal or stool culture tests

FMT stool donor inclusion criteria:

* Able to provide informed consent
* Able to complete donor screening
* Able to adhere to FMT stool collection and testing procedures

Renal transplant patient exclusion criteria:

* Still in hospital at week 7 following organ transplantation
* Pregnant or planning to become pregnant
* Breastfeeding
* Participating in another interventional or investigational study
* Neutropenic (ANC < 0.5)
* Presence of colostomy or ileostomy
* Has an active intestinal infection
* Fever > 38.0 or white blood count (WBC) count > 15,000
* Are taking a non-dietary probiotic supplement
* Require or are expected to require systemic antimicrobial therapy other than Pneumocystis prophylaxis or cytomegalovirus (CMV) therapy during the study period
* Has a severe underlying disease with anticipated survival less than 6 months
* Are unable to tolerate FMT or enema for any reason, or where their physician believes for any reason that FMT might pose a health risk to the subject
* Subjects who report a history of anaphylactoid food allergy will not be excluded but these allergies will be noted and donors will be required to avoid ingestion of these foods for at least three days prior to donation

FMT stool donor exclusion criteria:

* Presence of any of the following by stool examination: vancomycin-resistant Enterococci (VRE), Salmonella, Shigella, shiga toxin-producing E. coli, Yersinia, Campylobacter, extended spectrum beta-lactamase (ESBL) producing organisms or carbapenemase-producing Enterobacteriaceae (CRE), pathogenic ova or parasites, C. difficile toxin B (by PCR), or rotavirus, adenovirus and norovirus
* History of any type of active cancer aside from melanoma
* Risk factors for acquisition of HIV, syphilis, Hepatitis B, Hepatitis C, prion or any neurological disease as determined by the donor questionnaire
* History of gastrointestinal comorbidities, e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation or diarrhea, or colostomy or ileostomy
* Receipt of blood transfusion from a country other than Canada in the preceding 6 months
* Antibiotic use or any systemic immunosuppressive agents in the 3 months prior to stool donation
* Receipt of any live vaccine within 3 months prior to stool donation
* Any current or previous medical or psychosocial condition or behaviors which in the opinion of the investigator may pose risk to the recipients or the donor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The elimination of the target multi-drug resistant organism (MDRO), using culture and molecular test-based screening of recipient stool, at both the 14 and 30 days post-FMT. | 3 years

SECONDARY OUTCOMES:
Compare proportions, type and timing of adverse events post-FMT | 3 years
Proportions of recolonization over 180 days | 3 years
Timing of recolonization over 180 days | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Providence Health Care - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver Coastal Health - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided